CLINICAL TRIAL: NCT06650020
Title: The Impact of Synchronous Online Learning on the Theoretical Training of New Paediatric Nurses: A Prospective Randomized Trial
Brief Title: The Impact of Synchronous Online Learning on the Theoretical Training of New Paediatric Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-528
Record Dates: First submitted 2024-06-02; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Intervention
Keywords: Synchronous online learning; Randomized controlled trial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (Experimental): The control group adhered to the traditional offline model of centralized training
  Interventions: Other: the traditional offline model of centralized training
- synchronous online learning group (Experimental): The experimental group implemented an online training modality.
  Interventions: Other: synchronous online learning

INTERVENTIONS:
Other: synchronous online learning — Each participant in this cohort selected a suitable and peaceful learning environment, characterized by ample lighting and strong network connectivity. Equipped with laptops, participants logged into the Tencet conference software ten minutes prior to the session, entered their authentic names, completed the sign-in process five minutes before the course started, and kept their cameras activated throughout the session. During the instructional phase, both the teacher and control group were physically present. While the teacher instructed the control group, screen sharing through Tencet conference software allowed trainees in the experimental group to have clear visual access to instructional materials while audibly receiving instruction through microphones.
  Arms: synchronous online learning group
Other: the traditional offline model of centralized training — The control group adhered to the traditional offline model of centralized training, which involved a training facility spanning 100 square meters and accommodating seating for 150 participants. The front section of the training room was equipped with various amenities, such as a projection screen, podium, computer, and microphone, all available for use by the instructors. Throughout the training period, the lecturer provided in-person instruction on-site, allowing trainees to engage in real-time interaction by raising their queries.
  Arms: the control group

SUMMARY:
To examine the impact of synchronous online learning on the effectiveness of theoretical training and self-efficacy among newly graduated pediatric nurses.We carried out a Prospective randomized controlled trial.The sample comprised 45 newly graduated pediatric nurses randomly assigned to an experimental cohort group or a cohort group.The control group underwent traditional face-to-face teaching, whereas the experimental group engaged in synchronous online learning.Comparative analysis encompassed the test score from post-session 10-minute assessments, evaluations conducted after one week, and those after one month, alongside their academic self-efficacy scores.

DETAILED DESCRIPTION:
Aims To examine the impact of synchronous online learning on the effectiveness of theoretical training and self-efficacy among newly graduated pediatric nurses.

Design Prospective randomized controlled trial. Methods The sample comprised 45 newly graduated pediatric nurses randomly assigned to an experimental cohort group or a cohort group.The control group underwent traditional face-to-face teaching, whereas the experimental group engaged in synchronous online learning.Comparative analysis encompassed the test score from post-session 10-minute assessments, evaluations conducted after one week, and those after one month, alongside their academic self-efficacy scores.

ELIGIBILITY:
Inclusion Criteria:

1. Novice pediatric nurses
2. Continued engagement in full-time nursing studies;
3. Successful completion of pre-employment training evaluation at the hospital.

Exclusion Criteria:

1. Inability to complete all specified training modules;
2. Unwillingness to participate in the study.

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Theoretical Evaluation Scores | The assessment occurred across multiple stages: the pre-class test, the 10-minute post-class test, one week, and one month.
  The examination paper was an internally developed document, with the instructor independently formulating the topics relevant to the course. The content was carefully aligned with the course's instructional material and underwent rigorous review by the teaching team. Each unit of course content was accompanied by five corresponding questions, including two single-choice, two multiple-choice, and one judgement-based query. Overall, the examination comprised 60 questions, each worth 2 points, resulting in a total of 120 points.

SECONDARY OUTCOMES:
Scores of Academic Self-efficacy | one month
  The evaluation questionnaire was divided into two domains: learning aptitude self-efficacy and learning behavioral self-efficacy, comprising a total of 22 test items. Learning aptitude self-efficacy refers to an individual's assessment and confidence in their ability to effectively navigate their studies, achieve commendable outcomes, and avoid academic shortcomings. On the other hand, learning behavioral self-efficacy focuses on an individual's evaluation and confidence in "relatively agree" earning 4 points, and "completely agree" earning 5 points. Within this structure, questions 14, 16, 17, and 20 are subject to reversed scoring. A higher cumulative score indicates increased academic self-efficacy. The combined total of the two dimensions represents the overall academic self-efficacy score. Similarly, a higher score indicates a heightened level of self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Hu, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China